CLINICAL TRIAL: NCT06049654
Title: Clinical Trial of the Results of Allegra vs Sapien Transcatheter Aortic Valves in Valve-In-Valve Indication
Brief Title: Comparison of Allegra vs Sapien Transcatheter Aortic Valves in Valve-In-Valve Indication
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación EPIC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EPIC34-VIVALL 2 TRIAL
Record Dates: First submitted 2023-08-17; First posted 2023-09-22 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Aortic Valve Stenosis; Structural Valve Deterioration
Keywords: Valve-In-Valve; Aortic stenosis; Aortic regurgitation; Trans-catheter aortic valve; Degenerated aortic valve
MeSH Terms: conditions — Aortic Valve Stenosis; Aortic Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVT ALLEGRA System TF (Active Comparator): NVT ALLEGRA System TF
  Interventions: Device: NVT ALLEGRA TAVI System TF
- EDWARDS SAPIEN 3 or SAPIEN ULTRA SYSTEM (Experimental): EDWARDS SAPIEN 3 or SAPIEN ULTRA SYSTEM
  Interventions: Device: EDWARDS SAPIEN 3 or SAPIEN ULTRA SYSTEM

INTERVENTIONS:
Device: NVT ALLEGRA TAVI System TF — Transcatheter aortic valve implantation of a NVT ALLEGRA TAVI System TF in patients with severe haemodynamical valve deterioration of a biological aortic valve implanted surgically
  Arms: NVT ALLEGRA System TF
Device: EDWARDS SAPIEN 3 or SAPIEN ULTRA SYSTEM — Transcatheter aortic valve implantation of an EDWARDS SAPIEN 3 SYSTEM in patients with severe haemodynamical valve deterioration of a biological aortic valve implanted surgically
  Arms: EDWARDS SAPIEN 3 or SAPIEN ULTRA SYSTEM

SUMMARY:
The VIVALL-2 study is a randomized trial to compare the self-expandable supra-annular Allegra and the balloon-expandable intra-annular Edwards transcatheter valve systems in patients with degenerated biological aortic surgical valve.

DETAILED DESCRIPTION:
In the VIVALL.2 study, 104 patients with severely degenerated biological aortic surgical valve accepted for vave-in-valve procedure (transcatheter aortic valve implantation) will be randomized to be treated with the self-expandable supra-annular Allegra or the balloon-expandable intra-annular Edwards systems. The primary end-point will be trans-aortic mean gradient determined by trans-thoracic echocardiography at 30 days. The proportion of patients with moderate or severe prosthesis mismatch at 30 days will be a secondary end-.point. Different countries will participate in the study.

ELIGIBILITY:
Inclusion Criteria:

Patients meeting ALL the following criteria will be included:

* Patients aged ≥ 18 years.
* Severe haemodynamical valve deterioration of a biological aortic valve implanted surgically, including severe valve stenosis (effective aortic valve area < 1.0 cm2) and/or severe valve regurgitation.
* The patient has cardiac symptoms and/or deterioration of left ventricular ejection fraction attributable to the aortic valve disease.
* Heart team decision of VIV procedure.
* Patient is willing to return at 30 days for TTE and to be clinically contacted at 1 year.

Exclusion Criteria:

Patients meeting, at least, 1 of the following criteria will be excluded:

* Patients who openly express their refusal to participate in the study.
* Female patients in gestational age.
* Presence or suspicious of biological aortic valve thrombosis.
* Known hypersensitivity or contraindication to antithrombotic therapy (or inability to be anticoagulated during the procedure), nitinol, or sensitivity to contrast media which cannot be adequately pre-medicated.
* Ongoing sepsis and/or suspicious or diagnosis of endocarditis.
* Patients whose life expectancy is < 1 year due to non-cardiac comorbid conditions.
* Medical, social, or psychological conditions that preclude the subject from appropriate consent or adherence to the protocol required follow-up exams.
* True inner diameter of the prosthetic valve > 27 mm.
* Transfemoral access inadequate to accommodate an 18F sheath.
* Patients included in other clinical trials (excluding registries).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Trans-aortic mean gradient after Valve-in-Valve procedure, measured by transthoracic echocardiography (TTE). | 30 days
  Trans-aortic mean gradient after Valve-in-Valve procedure, measured by transthoracic echocardiography (TTE).

SECONDARY OUTCOMES:
Proportion of patients with device success after the Valve In Valve (VIV) procedure | 30 days
  Device success after the VIV procedure to the VARC-3 criteria
Proportion of patients with a trans-aortic mean gradient higher than 20 mmHg after the VIV procedure | 30 days
  Proportion of patients with a trans-aortic mean gradient higher than 20 mmHg after the VIV procedure
Proportion of patients with moderate or severe prosthesis mismatch 30 days after the VIV intervention. | 30 days
  Proportion of patients with moderate or severe prosthesis mismatch 30 days after the VIV intervention.
Early safety at 30 days as defined by Valve Academic Research Consortium 3 (VARC-3) criteria | 30 days
  freedom from: all-cause mortality, all stroke, VARC type 2-4 bleeding, major vascular, access-related, or cardiac structural complication, acute kidney injury stage 3 or 4, moderate or severe aortic regurgitation, new permanent pacemaker due to procedure related conduction abnormalities, surgery or intervention related to the device.
Clinical efficacy at 1 year as defined by VARC-3 criteria | 1 year
  freedom from: all-cause mortality, all stroke, hospitalization for procedure- or valve related causes, KCCQ Overall Summary Score <45 or decline from baseline of >10 point.
Trans-aortic mean gradient | 1 year
  Trans-aortic mean gradient 1 year after TAVR procedure
Death | 1 year
  Incidence of Death
Stroke | 1 year
  Incidence of Stroke

CONTACTS AND LOCATIONS:
Locations (9):
- Spain (6):
  - Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de La Paz, Madrid
  - Hospital Universitario Puerta De Hierro, Majadahonda
  - Hospital Clínico Universitario de Salamanca, Salamanca
  - Hospital Universitari I Politècnic de La Fe, Valencia
- United Kingdom (3):
  - Manchester University NHS Foundation Trust, Manchester
  - Freeman Hospital, Newcastle
  - Morriston Hospital, Swansea, Swansea

REFERENCES:
- [Background] Moreno R, Baz JA, Moreu J, Berenguer A, Gonzalvez-Garcia A, Galeote G, Hernandez U, Canton T, Jimenez-Valero S, Jurado-Roman A, Moya H, Lazaro E. Transcatheter aortic valve implantation for degenerated aortic valves: Experience with a new supra-annular device. The Spanish Allegra valve-in-valve (SAVIV) registry. Catheter Cardiovasc Interv. 2021 Aug 1;98(2):365-370. doi: 10.1002/ccd.29742. Epub 2021 Apr 23. PMID 33890713
- [Background] Hirji SA, Percy ED, Zogg CK, Malarczyk A, Harloff MT, Yazdchi F, Kaneko T. Comparison of in-hospital outcomes and readmissions for valve-in-valve transcatheter aortic valve replacement vs. reoperative surgical aortic valve replacement: a contemporary assessment of real-world outcomes. Eur Heart J. 2020 Aug 1;41(29):2747-2755. doi: 10.1093/eurheartj/ehaa252. PMID 32445575
- [Background] Bleiziffer S, Simonato M, Webb JG, Rodes-Cabau J, Pibarot P, Kornowski R, Windecker S, Erlebach M, Duncan A, Seiffert M, Unbehaun A, Frerker C, Conzelmann L, Wijeysundera H, Kim WK, Montorfano M, Latib A, Tchetche D, Allali A, Abdel-Wahab M, Orvin K, Stortecky S, Nissen H, Holzamer A, Urena M, Testa L, Agrifoglio M, Whisenant B, Sathananthan J, Napodano M, Landi A, Fiorina C, Zittermann A, Veulemans V, Sinning JM, Saia F, Brecker S, Presbitero P, De Backer O, Sondergaard L, Bruschi G, Franco LN, Petronio AS, Barbanti M, Cerillo A, Spargias K, Schofer J, Cohen M, Munoz-Garcia A, Finkelstein A, Adam M, Serra V, Teles RC, Champagnac D, Iadanza A, Chodor P, Eggebrecht H, Welsh R, Caixeta A, Salizzoni S, Dager A, Auffret V, Cheema A, Ubben T, Ancona M, Rudolph T, Gummert J, Tseng E, Noble S, Bunc M, Roberts D, Kass M, Gupta A, Leon MB, Dvir D. Long-term outcomes after transcatheter aortic valve implantation in failed bioprosthetic valves. Eur Heart J. 2020 Aug 1;41(29):2731-2742. doi: 10.1093/eurheartj/ehaa544. PMID 32592401
- [Background] Rodes-Cabau J, Abbas AE, Serra V, Vilalta V, Nombela-Franco L, Regueiro A, Al-Azizi KM, Iskander A, Conradi L, Forcillo J, Lilly S, Calabuig A, Fernandez-Nofrerias E, Mohammadi S, Panagides V, Pelletier-Beaumont E, Pibarot P. Balloon- vs Self-Expanding Valve Systems for Failed Small Surgical Aortic Valve Bioprostheses. J Am Coll Cardiol. 2022 Aug 16;80(7):681-693. doi: 10.1016/j.jacc.2022.05.005. Epub 2022 May 18. PMID 35597385
- [Background] Hahn RT, Webb J, Pibarot P, Ternacle J, Herrmann HC, Suri RM, Dvir D, Leipsic J, Blanke P, Jaber WA, Kodali S, Kapadia S, Makkar R, Thourani V, Williams M, Salaun E, Vincent F, Xu K, Leon MB, Mack M. 5-Year Follow-Up From the PARTNER 2 Aortic Valve-in-Valve Registry for Degenerated Aortic Surgical Bioprostheses. JACC Cardiovasc Interv. 2022 Apr 11;15(7):698-708. doi: 10.1016/j.jcin.2022.02.014. PMID 35393102
- [Background] Sa MPBO, Van den Eynde J, Simonato M, Cavalcanti LRP, Doulamis IP, Weixler V, Kampaktsis PN, Gallo M, Laforgia PL, Zhigalov K, Ruhparwar A, Weymann A, Pibarot P, Clavel MA. Valve-in-Valve Transcatheter Aortic Valve Replacement Versus Redo Surgical Aortic Valve Replacement: An Updated Meta-Analysis. JACC Cardiovasc Interv. 2021 Jan 25;14(2):211-220. doi: 10.1016/j.jcin.2020.10.020. PMID 33478639
- [Background] Landes U, Sathananthan J, Witberg G, De Backer O, Sondergaard L, Abdel-Wahab M, Holzhey D, Kim WK, Hamm C, Buzzatti N, Montorfano M, Ludwig S, Conradi L, Seiffert M, Guerrero M, El Sabbagh A, Rodes-Cabau J, Guimaraes L, Codner P, Okuno T, Pilgrim T, Fiorina C, Colombo A, Mangieri A, Eltchaninoff H, Nombela-Franco L, Van Wiechen MPH, Van Mieghem NM, Tchetche D, Schoels WH, Kullmer M, Tamburino C, Sinning JM, Al-Kassou B, Perlman GY, Danenberg H, Ielasi A, Fraccaro C, Tarantini G, De Marco F, Redwood SR, Lisko JC, Babaliaros VC, Laine M, Nerla R, Castriota F, Finkelstein A, Loewenstein I, Eitan A, Jaffe R, Ruile P, Neumann FJ, Piazza N, Alosaimi H, Sievert H, Sievert K, Russo M, Andreas M, Bunc M, Latib A, Godfrey R, Hildick-Smith D, Chuang MA, Blanke P, Leipsic J, Wood DA, Nazif TM, Kodali S, Barbanti M, Kornowski R, Leon MB, Webb JG. Transcatheter Replacement of Transcatheter Versus Surgically Implanted Aortic Valve Bioprostheses. J Am Coll Cardiol. 2021 Jan 5;77(1):1-14. doi: 10.1016/j.jacc.2020.10.053. PMID 33413929